CLINICAL TRIAL: NCT00000932
Title: A Prospective Study of Long-Term Clinical, Virologic, and Immunologic Outcomes in HIV-Infected Individuals
Brief Title: A Study of the Long-Term Outcomes of HIV-Positive Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: CPCRA 060; 10110 (Registry Identifier: DAIDS ES number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: HIV Infections
Keywords: Prospective Studies; HIV-1; Drug Therapy, Combination; Drug Resistance, Microbial; CD4 Lymphocyte Count; Disease Progression; Treatment Outcome; Genotype; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- A: Participants currently enrolled in or currently being followed in an ongoing qualifying study. Qualifying studies can be found in the protocol.
- B: Participants previously enrolled in but not currently being followed in a qualifying study. Qualifying studies can be found in the protocol.
- C: Antiretroviral-naive participants not enrolling in a qualifying study (i.e., patients starting treatment outside the first study or patients deferring treatment)

SUMMARY:
The purpose of this study is to collect information about life spans and HIV-related illnesses in multiple groups of HIV-positive patients with varying anti-HIV treatment experience, including no treatment at all.

Anti-HIV treatment has been successful in slowing disease progression in many patients. However, there are still questions regarding the best way to use anti-HIV drugs. This study is designed to provide long-term monitoring of patients who have already received anti-HIV treatment as well as patients who are just beginning treatment or have decided not to receive treatment.

DETAILED DESCRIPTION:
Highly active antiretroviral therapy (HAART) often results in short-term benefits for people with HIV in terms of reduced plasma viral levels and increased CD4 cell counts. When used at an early stage of HIV disease, however, the clinical benefit of HAART is uncertain. Many questions still remain regarding the optimal use of antiretroviral therapies, such as the timing of initial antiretroviral therapy and the composition of the best combination regimen to use initially or after virologic failure. Randomized trials of different starting antiretroviral regimens (e.g., FIRST [CPCRA 058]), different regimens after initial virologic failure (e.g., PIP [CPCRA 057]), and different management strategies for HIV infection (e.g., bis-POM [CPCRA 039], NvR [CPCRA 042], GART [CPCRA 046], and IL-2 VL/Dose [CPCRA 059] are being conducted by the CPCRA. [AS PER AMENDMENT 2/28/01: The MDR-HIV (CPCRA 064) protocol is now included as an example of a different management strategy for HIV infection, whereas the bis-POM (CPCRA 039) protocol is no longer included.] This study provides a mechanism for long-term monitoring of patients enrolled in these trials as well as antiretroviral-naive patients who are either starting treatment or electing to defer treatment.

Patients are divided into 3 groups. Group A consists of patients currently enrolled in or currently being followed in an ongoing qualifying study (see Purpose for CPCRA trials which qualify). Group B consists of patients previously enrolled in but not currently being followed in a qualifying study. Group C consists of antiretroviral-naive patients not enrolling in a qualifying study (i.e., patients starting treatment outside the FIRST study or patients deferring treatment). Patients in Group A undergo monitoring of selected clinical and laboratory parameters (including plasma HIV RNA levels and CD4 cell counts) once every 4 weeks beginning after completion of all follow-up appointments for all other protocols in which they were enrolled. Patients in Groups B and C undergo monitoring of selected clinical and laboratory parameters (including plasma HIV RNA levels and CD4 cell counts) once every 4 months. Patients are followed for at least 5 years. [AS PER AMENDMENT 2/28/01: Patients who are not being followed in a qualifying protocol and are antiretroviral naive at enrollment or were previously enrolled in the FIRST (CPCRA 058) protocol undergo blood draws at enrollment and then annually for measurement of plasma HIV levels by a CPCRA-approved laboratory and future CPCRA-approved, HIV-related research. Patients who relocate to a non-CPCRA affiliated site are asked to sign a consent for ongoing release (every 4 months) of their medical records from their new health care provider to the CPCRA.]

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are 13 years of age or older (consent of parent or guardian required if under the age of 18).
* Are HIV-positive.
* Have either: (1) no previous experience with anti-HIV treatment (defined as no previous protease inhibitor or nonnucleoside reverse transcriptase inhibitor use, 1 week or less of lamivudine use, and 4 weeks or less of cumulative nucleoside reverse transcriptase inhibitor use) or (2) current or previous enrollment in a qualifying CPCRA study.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV infected individuals
Sampling Method: Probability Sample
Enrollment: 3669 (Actual)
Dates: Start 1999-03; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Clinical disease progression or death | Throughout study

SECONDARY OUTCOMES:
Survival | Throughout study
Selected metabolic, hepatic, and cardiovascular conditions | Throughout study
Changes in viral load | Throughout study
Changes in CD4 count | Throughout study
Changes in HIV treatment methods | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Jay Kostman, Study Chair; Roberta Luskin-Hawk, Study Chair
Locations (91):
- United States (91):
  - Dr. M. Estes Med. Practice CRS, Mill Valley, California
  - Dr. Robert Scott Med. Practice CRS, Oakland, California
  - East Bay AIDS Ctr. CRS, Oakland, California
  - Dr. Shawn Hassler Med. Practice CRS, San Francisco, California
  - Positive Health Program Clinic (San Francisco Gen. Hosp.) CRS, San Francisco, California
  - Dr. Virginia Cafaro Med. Practice CRS, San Francisco, California
  - Dr. William Owen Med. Practice CRS, San Francisco, California
  - Castro-Mission Health Ctr. CRS, San Francisco, California
  - Dr. Martin Mass Med. Practice CRS, San Francisco, California
  - St. Mary's Med. Ctr. of San Francisco CRS, San Francisco, California
  - San Francisco VAMC, Infectious Diseases Clinic CRS, San Francisco, California
  - UCSF PHP, Gen. Internal Medicine Practice CRS, San Francisco, California
  - Beacon Clinic at Boulder CRS, Boulder, Colorado
  - Denver Infectious Diseases Consultants CRS, Denver, Colorado
  - Kaiser Permanente of Denver CRS, Denver, Colorado
  - Univ. of Colorado Health Science Ctr. CRS, Denver, Colorado
  - Denver Public Health CRS, Denver, Colorado
  - Eastside Family Health Ctr. CRS, Denver, Colorado
  - APEX Family Medicine CRS, Denver, Colorado
  - South Denver Infectious Diseases Specialists, Accord Med. Ctr. CRS, Denver, Colorado
  - Denver Public Health CRS - INSIGHT, Denver, Colorado
  - Western Infectious Disease Consultants CRS, Wheat Ridge, Colorado
  - Univ. of Connecticut Health Ctr. CRS, Farmington, Connecticut
  - Yale Univ. School of Medicine, NE ProACT - New Haven CRS, New Haven, Connecticut
  - Hosp. of St. Raphael CRS, New Haven, Connecticut
  - Dotson & Hodge Med. Group, L.L.C. CRS, Washington D.C., District of Columbia
  - Dr. Timothy A. Price Med. Practice CRS, Washington D.C., District of Columbia
  - Washington DC VAMC, Washington Regional AIDS Program, Infectious Diseases CRS, Washington D.C., District of Columbia
  - Klein & Slotten Medical Associates CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr. INSIGHT CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Univ. of Illinois Family Ctr. for Infectious Disease CRS, Chicago, Illinois
  - Lakeshore Infectious Disease Associates CRS, Chicago, Illinois
  - North Side Family Medicine CRS, Chicago, Illinois
  - Northwestern Memorial Physicians Group CRS, Chicago, Illinois
  - Triad Health Practice/Ill. Masonic Med. Ctr. CRS, Chicago, Illinois
  - Earl K. Long Med. Ctr., LSU - Mid City EIC Clinic CRS, Baton Rouge, Louisiana
  - James Osterberger, MD (Private Med. Practice) CRS, Baton Rouge, Louisiana
  - Med. Ctr. of Louisiana at New Orleans, HIV Outpatient Clinics CRS, New Orleans, Louisiana
  - Tulane University Health Sciences Center, Louisiana Community AIDS Research Program(LaCARP) CRS, New Orleans, Louisiana
  - Memorial Med. Ctr., Hematology-Oncology Services CRS, New Orleans, Louisiana
  - New Orleans VAMC CRS, New Orleans, Louisiana
  - CRI-Boston CRS, Boston, Massachusetts
  - CRI-Springfield CRS, Springfield, Massachusetts
  - Harper Hosp., Detroit CRS, Detroit, Michigan
  - Wayne State Univ. INSIGHT CRS, Detroit, Michigan
  - Henry Ford Hosp. CRS, Detroit, Michigan
  - Detroit Community Health Connection, Inc. CRS, Detroit, Michigan
  - Detroit Community Health Connection-2 CRS, Detroit, Michigan
  - Cooper Univ. Hosp. CRS, Camden, New Jersey
  - ID Care Inc. - Hillsborough CRS, Hillsborough, New Jersey
  - Jersey Shore Univ. Med. Ctr. CRS, Neptune City, New Jersey
  - Cathedral Healthcare System, St. Michael's Med. Ctr. CRS, Newark, New Jersey
  - New Jersey Community Research Initiative, Jeffrey Bomser Clinic CRS, Newark, New Jersey
  - St. Joseph's Hosp. & Med. Ctr. of New Jersey CRS, Paterson, New Jersey
  - Raritan Bay Med. Ctr., Perth Amboy Division CRS, Perth Amboy, New Jersey
  - ID Care - Randolph CRS, Randolph Township, New Jersey
  - Infectious Disease Specialists of N.J., North Jersey Community Research Initiative CRS, Union, New Jersey
  - The Early Intervention Program at Kennedy Hosp. CRS, Voorhees Township, New Jersey
  - St. Vincent Hosp. & Med. Ctr. CRS, New York, New York
  - HHC Methadone Maintenance, Treatment Program Unit 1 CRS, New York, New York
  - Harlem Hospital Ctr./Columbia University CRS (Gordin CTU), New York, New York
  - Bronx Prevention Center CRS, The Bronx, New York
  - Bronx-Lebanon Hosp. Ctr. CRS, The Bronx, New York
  - Jacobi Med. Ctr., Ambulatory Care Pavillion CRS, The Bronx, New York
  - Jacobi Med. Ctr., The Bronx, New York
  - Montefiore Med. Ctr., AIDS Ctr. CRS, The Bronx, New York
  - Multnomah County Health Dept., HIV Health Services Ctr. CRS, Portland, Oregon
  - Legacy Clinic Good Samaritan CRS, Portland, Oregon
  - The Research & Education Group-Portland CRS, Portland, Oregon
  - Providence Portland Med. Ctr., Ambulatory Care and Education Ctr. CRS, Portland, Oregon
  - Kaiser Immune Deficiency Clinic of Portland CRS, Portland, Oregon
  - Legacy Clinic Emanuel CRS, Portland, Oregon
  - Oregon Health & Sciences Univ. Internal Medicine (L-475) CRS, Portland, Oregon
  - Salem Hosp. CRS, Salem, Oregon
  - Kaiser Permanente Lancaster Clinic CRS, Salem, Oregon
  - Philadelphia FIGHT - Dr. Jay Kostman CRS, Philadelphia, Pennsylvania
  - Temple Univ. School of Medicine CRS, Philadelphia, Pennsylvania
  - Legacy Community Health Services, Inc. CRS, Houston, Texas
  - Baylor College of Medicine, Thomas St. Clinic CRS, Houston, Texas
  - Houston AIDS Research Team CRS, Houston, Texas
  - Michael E. DeBakey VAMC CRS, Houston, Texas
  - Thomas Street Clinic CRS, Houston, Texas
  - Hanover Med. Park (Mechanicsville, VA) CRS, Mechanicsville, Virginia
  - Eastern Virginia Med. School, Ctr. for the Comprehensive Care of Immune Deficiency CRS, Norfolk, Virginia
  - Petersburg Health Care Alliance CRS, Petersburg, Virginia
  - CrossOver Health Ctr. CRS, Richmond, Virginia
  - South Richmond Health Care Ctr. CRS, Richmond, Virginia
  - Hunter Holmes McGuire VAMC CRS, Richmond, Virginia
  - VCU Health Systems, Infectious Disease Clinic CRS, Richmond, Virginia
  - Virginia Commonwealth Univ. Medical Ctr. CRS, Richmond, Virginia

REFERENCES:
- [Result] Goetz MB, Leduc R, Kostman JR, Labriola AM, Lie Y, Weidler J, Coakley E, Bates M, Luskin-Hawk R; Long-Term Monitoring Study (CPCRA 060) and Terry Beirn Community Programs for Clinical Research on AIDS (CPCRA). Relationship between HIV coreceptor tropism and disease progression in persons with untreated chronic HIV infection. J Acquir Immune Defic Syndr. 2009 Mar 1;50(3):259-66. doi: 10.1097/QAI.0b013e3181989a8b. PMID 19194318